CLINICAL TRIAL: NCT03483519
Title: Efficacy of Preoperative Muscle Training on Postoperative Recovery and Function in Patients Undergoing Total Hip or Knee Replacement
Brief Title: Efficacy of Preoperative Muscle Training on Postoperative Orthopaedic Surgery Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20150684
Record Dates: First submitted 2016-08-03; First posted 2018-03-30 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Arthroplasty; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Rehabilitation; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): Patients in the Prehabilitation Group and are randomized to the Experimental Group will undergo a 6 Week Exercise Program plus Standard of Care
  Interventions: Other: Rehabilitation
- Standard of Care (Active Comparator): Patients in the Standard of Care will not receive an additional an exercise program, patients will receive the usual care received by all orthopaedic patients.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Rehabilitation — Patients randomized to the Experimental Group will undergo a 6 Week Exercise Program plus Standard of Care
  Arms: Prehabilitation
Other: Standard of Care — Patients randomized to the Active Comparator Group will not undergo an exercise program, patients will receive the standard of care used at The Ottawa Hospital for hip and knee surgeries. Standard of care protocol will be explained by each individual surgeon.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to assess the effectiveness of a preoperative muscle training program on hip or knee TJA (Total Joint Arthroplasty). It aims to improve hospital discharge readiness and functional capacity in both the short and long-term. One of the key factors affecting recovery after TJA is how well the patient functions before their surgery. Thus, interventions addressing preoperative function are expected to be beneficial.

DETAILED DESCRIPTION:
Although total hip or knee joint replacement is beneficial in treating severe hip or knee osteoarthritis, a significant number of patients take longer to recover in the hospital or have a non-optimal quality of life after the surgery. These patients often have difficulties in accomplishing basic essential everyday tasks such as walking and stair climbing, both shortly and long after surgery. It has been previously shown through research that difficulties to do basic tasks before surgery delays recovery and negatively affects long-term function. It has also been shown that these difficulties are associated with reduced strength in hip or knee muscles present before surgery, caused by lack of activity of patients. This study will determine if a hip or knee muscle strengthening exercise program accomplished before surgery can improve hospital recovery, capacity to accomplish basic activities, and quality of life two days, six weeks and six months after joint replacement surgery. If this exercise program is shown to be beneficial, it will be easily used by patients when waiting for their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older undergoing unilateral total hip or knee arthroplasty due to osteoarthritis;
* WOMAC functional subscale less than 66.5/100.

Exclusion Criteria:

* Patients under 18 years of age;
* Patients undergoing joint revision on the affected side;
* patients under the same day discharge protocol;
* Patients undergoing bilateral arthroplasty;
* Patients suffering from other previously diagnosed lower-limb problems limiting their capacity to accomplish the exercise program;
* Patients having surgery in less than 16 weeks after verbal consent;
* Patients unable or unwilling to commit to required study follow-ups;
* Patients with no fixed address;
* Patients with a cognitive impairment that may preclude questionnaire completion;
* Pregnant or suspected pregnant women as dual-energy x-ray (DXA) used in this study may be harmful to a fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
HOOS or KOOS Questionnaire to assess self-reported pain | 12 months
  The Hip Disability and Osteoarthritis Outcome Score (HOOS) or Knee Injury and Osteoarthritis Outcome Score (KOOS). A standardized set of questions to assess the function of the hip or knee (dependent on which surgery the patient is undergoing). The KOOS/HOOS are comprised of 6 sections: 1) Symptoms (3 items), 2) Stiffness (2 items), 3) Pain (10 items), 4) Function Daily Living (17 items), 5) Function/Sports and Recreation (4 items), 6) Quality of Life (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.

SECONDARY OUTCOMES:
Timed-Up-and-Go (TUG) | 12 months
  Assesses the time that a patient takes to rise from a chair, walk three metres, turn around, walk back to the chair, and sit down. Time will be measured in seconds.
Timed Stair Test | 12 months
  Assesses the time that a patient takes to ascend and descend a flight of 10 stair, while holding on to the handrail. Time will be measured in seconds.
Length of hospital stay | 1 month
  Length of stay will be calculated from the date of surgery to discharge from an inpatient bed. Length of stay will be measured in days until hospital discharge.
Post-surgical Complications | 30 days
  Post-operative complications and adverse events will be collected using the Ottawa Hospital data warehouse coding data.
Hip or Knee Muscle Strength | 12 months
  For patients undergoing hip surgery, hip abductor strength will be assessed with a hand held dynamometer with the patient in the side-lying position. For patients undergoing knee surgery, quadriceps strength will be measured with a hand held dynamometer with the patient in the supine position and the knee flexed at 60 degrees. A dynamometer is a small machine hand-held by the research assistant that you push on with your leg in order to measure the strength of your muscle (measured in kilograms). The average of three trials will be used. Absolute (affected side only) and relative (difference between non-affected and affected side) strength values will be calculated. Muscle strength will be assessed at baseline, two weeks before surgery, six months and one year after surgery.
Muscle Mass measured with dual-energy x-ray absorptiometry | 12 months
  Body weight and height will be measured. A method called dual-energy x-ray (DXA) will also be used to measure bone density, percent fat and percent lean body mass. The patient will lie on an examination table, wearing a hospital gown, while a low-intensity x-ray will scan the entire body. The measurement takes approximately 20 minutes. The only risk is a minimal x-ray exposure of less than 0.003 mSv, which is less than the natural exposure to sunlight during the course of 1 day. Muscle mass will be assessed at baseline, two weeks before surgery, six months and one year after surgery.
Generic Health Status measured by the Questionnaire EQ-5D-5L | 12 months
  A standardized set of questions to assess generic health status. The EQ-5D-5L questionnaire consists of 2 pages: the EQ-5D descriptive system (5 items) and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The patient is asked to tick the box that is most appropriate to their health within the 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled as 100 ('The best health you can imagine) and 0 (The worst health you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, Principal Investigator — Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Sled EA, Khoja L, Deluzio KJ, Olney SJ, Culham EG. Effect of a home program of hip abductor exercises on knee joint loading, strength, function, and pain in people with knee osteoarthritis: a clinical trial. Phys Ther. 2010 Jun;90(6):895-904. doi: 10.2522/ptj.20090294. Epub 2010 Apr 8. PMID 20378679
- [Derived] Pacheco-Brousseau L, Dobransky J, Jane A, Beaule PE, Poitras S. Feasibility of a preoperative strengthening exercise program on postoperative function in patients undergoing hip or knee arthroplasty: a pilot randomized controlled trial. Pilot Feasibility Stud. 2022 Jul 30;8(1):162. doi: 10.1186/s40814-022-01126-9. PMID 35908037